CLINICAL TRIAL: NCT05021471
Title: Effects Of Stretching With And Without Pressure Biofeeback On Hamstring Muscle Flexibility In Patients With Postural Syndrome
Brief Title: Stretching With And Without Pressure Biofeeback In Patients With Postural Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0114 Hashim
Record Dates: First submitted 2021-08-23; First posted 2021-08-25 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Postural; Defect
Keywords: Pressure biofeedback unit,; Stretching Hamstring Muscles; Active Knee Extension Test
MeSH Terms: interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Twenty nine (29) patients will be treated stretching of hamstring with pressure biofeedback.
  Interventions: Other: biofeedback
- Group B (Active Comparator): Twenty nine (29) patients will be treated stretching of hamstring without pressure biofeedback.
  Interventions: Other: hamstrings stretching

INTERVENTIONS:
Other: biofeedback — Twenty nine (29) patients will be treated stretching of hamstring with pressure biofeedback.
  Arms: Group A
Other: hamstrings stretching — Twenty nine (29) patients will be treated stretching of hamstring without pressure biofeedback.
  Arms: Group B

SUMMARY:
Postural syndrome describes a variety of conditions in which repetitive or continued bad posture over a long period of time causes pain and reduced function in the muscles and joints.

Improper posture can cause pain throughout the length of the spine from the neck to the pelvis. Modern sedentary style of living is one of the main reasons for postural abnormalities evident in modern society. The prolonged sitting hours required in most of the jobs, and educational setups can affect flexibility of soft tissues, especially two joint muscles. Bad posture while standing or walking, if left uncorrected, can worsen over time and lead to pain and dysfunction. Hamstring is a key component of flexibility in the human body and it is more prone to get tightened. Many reasons can lead to the development of hamstring tightness such as genetic predisposition, injury to muscle, and adaptive shortening due to some chronic condition. Short hamstring muscles, because of their attachments to the posterior leg and to the ischial tuberosity, may limit hip flexion ROM and induces posterior pelvic tilt and decreased lumbar lordosis, which can result in LBP The purpose of this study will be to find out the effects of stretching with and without pressure biofeedback unit (PBU) on hamstring muscle flexibility in patients with postural syndrome. The active knee extension (AKE) test will be used to determine the length of the hamstring muscles using a goniometer. A PBU will be used to maintain the anterior pelvic tilt position during active knee extension (AKE) test or stretching, by monitoring the pressure of airbag. Patients will be recruited into study by convenient sampling technique after that will be allocated to groups by simple random assignment. All participants will actively stretch three days per week for four weeks. After collecting data from defined study setting, data will be entered and analyzed by using Statistical Package for the Social Sciences (SPSS) for Windows software, version 25.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of aged 18 to 25 years with hamstrings shortening less than 70 degrees are included in the study

Exclusion Criteria:

* Subjects with any past hamstring injury within last 2 years

  * Low back pain since past 3 months
  * Current or recent (last 3 months) participation in a specific program designed to lengthen the hamstrings are excluded

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
range of joint | 4 weeks
  universal goniometer as range increase it shows betterment
pain of patient | 4 weeks
  NPRS The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman Bashir, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, McClure PW, Pratt N. The effect of hamstring muscle stretching on standing posture and on lumbar and hip motions during forward bending. Phys Ther. 1996 Aug;76(8):836-45; discussion 845-9. doi: 10.1093/ptj/76.8.836. PMID 8710963
- [Background] Jandre Reis FJ, Macedo AR. Influence of Hamstring Tightness in Pelvic, Lumbar and Trunk Range of Motion in Low Back Pain and Asymptomatic Volunteers during Forward Bending. Asian Spine J. 2015 Aug;9(4):535-40. doi: 10.4184/asj.2015.9.4.535. Epub 2015 Jul 28. PMID 26240711
- [Background] May S, Nanche G, Pingle S. High frequency of McKenzie's postural syndrome in young population of non-care seeking individuals. J Man Manip Ther. 2011 Feb;19(1):48-54. doi: 10.1179/2042618610Y.0000000004. PMID 22294854
- [Background] Makhsous M, Lin F, Bankard J, Hendrix RW, Hepler M, Press J. Biomechanical effects of sitting with adjustable ischial and lumbar support on occupational low back pain: evaluation of sitting load and back muscle activity. BMC Musculoskelet Disord. 2009 Feb 5;10:17. doi: 10.1186/1471-2474-10-17. PMID 19193245